CLINICAL TRIAL: NCT06041230
Title: Comparison of the Efficiency of Extracorporeal Shock Wave Therapy and Ultrasound-Guided Ozone Injection in Patients With Chronic Plantar Fasciitis
Brief Title: Comparison of the Efficiency of ESWT and Ozone Injection in Patients With Chronic Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Berke Aras, Associate Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2-23-3838
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Plantar Fascitis
Keywords: ozone therapy; ESWT

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided ozone injection therapy (Active Comparator)
  Interventions: Device: Ozone Generator
- Extracorporeal shock wave therapy (Active Comparator)
  Interventions: Device: Extracorporeal shock wave therapy device

INTERVENTIONS:
Device: Ozone Generator — Ultrasound guided ozone therapy
  Arms: Ultrasound guided ozone injection therapy
Device: Extracorporeal shock wave therapy device — Extracorporeal shock wave therapy device
  Arms: Extracorporeal shock wave therapy

SUMMARY:
Extracorporeal Shock Wave Therapy (ESWT) is a conservative treatment method that has been widely used in musculoskeletal diseases in recent years. Its mechanism is to provide hyperstimulation and vascularity increase with the help of acoustic waves focused on a specific area, thus accelerating healing and reducing pain. This method, which is frequently used in plantar fasciitis, is frequently applied to patients whose symptoms persist despite first-line treatment strategies.

Ozone injections have been frequently used in musculoskeletal disorders in recent years and are mainly used in osteoarthritis, osteomyelitis, tendon, fascia and ligament injuries, vertebra and disc pathologies and neuropathic pain. Analgesic effect on musculoskeletal system (release of endorphins, activation of antinociceptive system, reduction of edema) anti-inflammatory effect (regulation of cytokine release, reduction of superoxide radicals, modulation of prostaglandin), regulation of local oxygenation and circulation, tissue repair (neutralization of preteolytic enzymes, fibroblast proliferation) and has an antimicrobial effect. Although it is also used in the treatment of plantar fasciitis, there are limited articles on this subject in the literature.

In our study, it was aimed to compare the effectiveness of ESWT and ozone injection therapy, which are two treatment strategies with regenerative action mechanisms, in patients with resistant plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Heel pain lasting longer than 3 months
* Localized pain and tenderness on palpation on the medial aspect of the calcaneal tuberosity when the ankle is fully dorsiflexed.
* In the first step of walking, >50 mm according to VAS. and description of pain
* Presence of plantar fasciitis typical findings on ultrasonography (thickening more than 4 mm in the proximal plantar fascia with changes in fibril pattern)
* Failure to respond to conservative treatment before (nonsteroidal anti-inflammatory drugs, stretching, heel cushion, shoe modifications, orthotics, cold, heat, taping, massage)

Exclusion Criteria:

* being under the age of 18
* Any skin lesions in the heel area
* Inflammatory, rheumatic arthritis
* Having a history of fracture, trauma or operation in the heel area
* Systemic infection or malignancy
* Having a pacemaker
* Local injection to the heel area in the last 6 months or use of topical or oral nonsteroidal anti-inflammatory drugs in the last 2 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | pre-treatment, immediately post-treatment and three months follow-up
  measurement for pain severity, It is a value between 0-100. "0" means no pain and "100" means maximum pain.

SECONDARY OUTCOMES:
plantar fascia thickness | pre-treatment, immediately post-treatment and three months follow-up
  sonographic measurement for plantar fascia
Foot Function İndex | pre-treatment, immediately post-treatment and three months follow-up
  measurements for foot function. An increase in the value indicates worse foot functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR